CLINICAL TRIAL: NCT03890926
Title: The Physical Dosimetry Study and Preliminary Clinical Results of 3D-printing Non Co-planar Template Assisted With CT-guidance for Iodine-125 Seed Brachytherapy in Pelvic Recurrent Rectum Carcinoma After Surgery and External Beam Radiotherapy, a Retrospective Study
Brief Title: The Physical Dosimetry Study and Preliminary Clinical Results of 3D-printing Non Co-planar Template Assisted With CT-guidance for Iodine-125 Seed Brachytherapy in Pelvic Recurrent Rectum Carcinoma After Surgery and External Beam Radiotherapy
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PekingUTH RT
Record Dates: First submitted 2019-03-09; First posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Rectum Cancer, Recurrent; Brachytherapy, Radioisotope
Keywords: Three-Dimensional Printing; Rectum Cancer, Recurrent; Radioactive Iodine-125 seed implantation
MeSH Terms: conditions — Rectal Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- radioactive Iodine-125 seed implantation: All enrolled patients received the intervention previously as a conventional treatment.
  Interventions: Radiation: radioactive Iodine-125 seed implantation under the guidance of 3D template

INTERVENTIONS:
Radiation: radioactive Iodine-125 seed implantation under the guidance of 3D template — 3D-PNCT assisted with CT-guidance for radioactive Iodine-125 seed brachytherapy is a conventional treatment for patients with local recurrent rectal carcinoma. Retrospective data on the effectiveness and adverse effects of the past radioactive Iodine-125 seed implantation is collected.

SUMMARY:
This study observes the efficacy and side effects of 3D-printing non co-planar template(3D-PNCT) assisted with CT-guidance for radioactive Iodine-125 seed(RIS) brachytherapy in pelvic recurrent rectum carcinoma retrospectively, and analyzes the influence of clinical and dosimetric factors on the outcomes.

DETAILED DESCRIPTION:
3D-PNCT assisted with CT-guidance for radioactive Iodine-125 seed brachytherapy is a conventional treatment in Peking University Third Hospital. Radioactive Iodine-125 seed brachytherapy is the implantation of Iodine-125 seed into tumors.The radioactive Iodine-125 seed can release low dose of irradiation persistently which kills tumors cell and causes less damage to normal tissue at the same time. 3D-printing non co-planar template is made individually which guides the implantation of Iodine-125 seed into the tumor and ensures the accuracy of the position.This study collects the data of patients with pelvic recurrent rectal carcinoma who underwent 3D-PNCT assisted with CT-guidance for radioactive Iodine-125 seed implantation from 2015 to 2018. We evaluate the dose that covers 90% target volume(D90),the volume that 100% prescription dose covers(V100) and other dosimetric parameters after the implantation. The efficacy and adverse effects were observed. Local control(LC) time and overall survival(OS) time are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* treated with 3D-printing non co-planar template assisted with CT-guidance for Iodine-125 seed brachytherapy in Peking University Third Hospital
* histological proven recurrent rectal cancer
* inoperable local recurrent cases
* previous external beam radiotherapy, incapable of re-irradiation
* expected life span>3 months

Exclusion Criteria:

* serious medical illness
* unable to tolerate anesthesia
* blood coagulation dysfunction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with local recurrent rectal carcinoma who were treated with 3D-printing non co-planar template assisted with CT-guidance for Iodine-125 seed brachytherapy as a conventional treatment in Peking University Third Hospital during December 2015 to December 2018
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Overall survival time | From date of implantation to the date of death from any cause or the date of last observation. The last follow-up timepoint is February 2019.
  The time from the date of implantation to the date of death from any cause or the date of last observation. Outcomes were followed up every 3 months after enrollment.
Local control time | From date of implantation to the date of recurrence of the implanted tumor or the date of last observation. The last follow-up timepoint is February 2019.
  The time from the date of implantation to the date of recurrence of the implanted tumor or the date of last observation. Outcomes were followed up every 3 months after enrollment.

SECONDARY OUTCOMES:
Pain relief rate | 3 months after the implantation. The last follow-up point is February 2019.
  Numerical rating scales(NRS) was used to evaluate the grade of pain. Grade 7-9 was defined as serve pain. Grade 4-6 was defined as moderate pain and grade 1-3 was defined as mild pain. The pain before and after the implantation was evaluated and the pain relief rate was measured.
Incidence of adverse events | From date of implantation to the date of death from any cause or the date of last observation. The last follow-up timepoint is February 2019.
  The adverse events were evaluated by the toxicity criteria of the Radiation Therapy Oncology Group (RTOG). The rate of each adverse event was measured.

CONTACTS AND LOCATIONS:
Overall Officials: junjie wang, Ph.D, Principal Investigator — Radiotherapy Department,Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: CSR
Time Frame: Data will be available within 6 months of the study completion.
Access Criteria: Data access requests will be reviewed by an external Independent Review Panel. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Wang Z, Lu J, Liu L, Liu T, Chen K, Liu F, Huang G. Clinical application of CT-guided (125)I seed interstitial implantation for local recurrent rectal carcinoma. Radiat Oncol. 2011 Oct 18;6:138. doi: 10.1186/1748-717X-6-138. PMID 22004599
- [Derived] Wang L, Wang H, Jiang Y, Ji Z, Guo F, Jiang P, Li X, Chen Y, Sun H, Fan J, Li W, Li X, Wang J. The efficacy and dosimetry analysis of CT-guided 125I seed implantation assisted with 3D-printing non-co-planar template in locally recurrent rectal cancer. Radiat Oncol. 2020 Jul 25;15(1):179. doi: 10.1186/s13014-020-01607-2. PMID 32711542